CLINICAL TRIAL: NCT05372835
Title: Effects of Hypochlorous Acid Mouthwash on Oral Bacteria in Patients With Periodontal Disease and Staphylococcus Aureus
Brief Title: Hypochlorous Acid Mouthwash, Oral Bacteria, and Staphylococcus Aureus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Ying-Chu Lin, Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KMUHIRB-F(I)-20200042
Record Dates: First submitted 2022-04-28; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Water

STUDY DESIGN:
Intervention Model Description: The volunteers of patients with and without periodontal disease were recruited in the same day. Patients with periodontal disease were randomized into mouthwash group and mouthwash plus periodontal flosser group. Patients without periodontal disease were recruited as the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants have no idea in the usage of mouthwash or water. Participant with and without periodontal disease was blinded for the laboratory determining total oral bacterial count in saliva samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mouthwash (Experimental): The 15 mL of commercially available La Chlogen mouthwash (Republic of China Patent No. M616466) was used for intervention to rinse in mouth for 5 minutes. The main ingredient in the mouthwash is low-concentration high-purity HOCl (100 ppm) solution.
  Interventions: Other: La Chlogen mouthwash
- mouthwash and periodontal flosser (Experimental): The 15 ml of commercially available La Chlogen mouthwash (Republic of China Patent No. M616466) in conjunction with the La Chlogen periodontal flosser (Republic of China Patent No. M590033) were used for intervention in the mouth for 5 minutes. The main ingredient in the mouthwash is low-concentration high-purity HOCl (100 ppm) solution.
  Interventions: Other: La Chlogen mouthwash and La Chlogen periodontal flosser
- control (Placebo Comparator): The pure water without HOCl chemical was applied in this intervention to rinse in mouth for 5 minutes.
  Interventions: Other: water

INTERVENTIONS:
Other: La Chlogen mouthwash — Patients with periodontal disease were randomized into mouthwash group. Before the intervention, participants were asked to rinse 5 ml of water to deplete the food debris and the other residues. After this, the intervention was asked participants to rinse the commercially available La Chlogen mouthwash in mouth without spitting. After 5 minutes, the participants spit out the liquid, and the saliva samples were collected for further analysis.
  Arms: mouthwash
Other: water — Patients without periodontal disease were selected as a control group. Before the intervention, participants were asked to rinse 5 ml of water to deplete the food debris and the other residues. After this, the intervention was asked participants to rinse the pure water in mouth without spitting. After 5 minutes, the participants spit out the liquid, and the saliva samples were collected for further analysis.
  Arms: control
Other: La Chlogen mouthwash and La Chlogen periodontal flosser — Patients with periodontal disease were randomized into mouthwash and periodontal flosser group. Before the intervention, participants were asked to rinse 5 ml of water to deplete the food debris and the other residues. After this, the La Chlogen mouthwash in conjunction with the La Chlogen periodontal flosser were applied in mouth without spitting for interventions. After 5 minutes, the participants spit out the liquid, and the saliva samples were collected for further analysis.
  Arms: mouthwash and periodontal flosser

SUMMARY:
Mouthwash is one method of maintain oral health and to reduce the dental plaque and gum inflammation. However, the effects of mouthwash on oral bacteria were not consistent among different brands of them. The aims of present study were to determine the effects of a new designed mouthwash with hypochlorous acid on oral bacteria and Staphylococcus aureus. All participants were invited as a volunteer to attend this study from a private dental clinic and diagnosed by the same dentist. Patients with periodontal diseases were randomized selected as mouthwash group and mouthwash plus dental flossing device (La Chlogen, Taiwan) group. Patients for regular dental visit and without periodontal disease were invited as a control group having mouth rinse with water. After the inform consent was signed, participants completed the intervention study, saliva collection, and a simple survey under the guide of a dental assistant. Saliva samples were collected before and after the intervention for bacterial DNA extraction. A real-time polymerase chain reaction and S. aureus with serial dilutions were applied for the estimation of total oral bacterial count (TOBC) in saliva. An in vitro assay with CCK-8 reagent was apply to test the antibacterial ability of mouthwash.

DETAILED DESCRIPTION:
Finally there were 83 person recruited into the present study. A total of 53 patients with periodontal disease diagnosed by a periodontist, who were randomly assigned to the mouthwash-only group (26 patients) or the mouthwash plus periodontal flosser group (27 patients). There were 30 controls recruited into the present study. For the determination of oral bacterial counts, a real-time polymerase chain reaction and a pure strain of Staphylococcus aureus with a serial dilutions were applied to create a standardized growth curve for the estimation of oral bacterial counts in saliva. Before the intervention, participants were asked to rinse 5 ml of water to deplete the food debris and the other residues in mouth. The intervention was asked participants to rinse the 15 ml mouthwash or water for 5 minutes in oral cavity.

Participants were asked their health history and use of dental cleaning tools. The participants underwent relevant oral health examinations, and their oral health indices were also recorded. The mouthwash used for intervention in the present study was the 15 mL of commercially available La Chlogen mouthwash (Republic of China Patent No. M616466) for 5 minites. The main ingredient in the mouthwash is low-concentration high-purity HOCl (100 ppm). The HOCl solutions can be also used in conjunction with the La Chlogen periodontal flosser (Republic of China Patent No. M590033). The controls were instructed to gargle with pure water (15 ml) for 5 minutes. Each participant first underwent a pretest, in which after the participants' saliva samples were collected, their total oral bacterial count (TOBC) were measured. Thereafter, each participant rinsed their mouth with their assigned liquid (mouthwash, mouthwash plus periodontal flosser or water) without spitting. After 5 minutes, the participants spit out the liquid, and these saliva samples were collected and tested to determine the TOBC.

Each participant underwent two saliva sample collection sessions: pretest and posttest. Before the saliva collection, participant rinsed with 5 ml of water. After this, participants were asked to expectorate over a maximum period of 3 minutes into a 50 ml sterile centrifugation tube (Creative Biotechnology Co., Ltd., Taiwan) for the collection of unstimulated whole saliva. The collected specimen was then immediately placed in a portable ice box for storage, returned to the laboratory for the same-day bacterial DNA extraction. The saliva volume and weight of each sample was also recorded before the bacterial genomic DNA extraction process.

TOBC analysis: After the extraction of the bacterial genomic DNA, The real-time polymerase chain reaction (RT-PCR) techniques were used to quantify the total counts of oral bacteria in the saliva samples. Saliva sample was centrifuged at 2500 rpm for 5 minutes. The pellet was suspended with 300µl lysozyme solution (2.5 mg/mL). After being mixed evenly, the mixture was transferred into a 1.5mL eppendorf tube and placed on ice for 1 hour. Thereafter, 10% SDS (20µL), 0.5M EDTA (80µL), and 20mg/mL proteinase K (10µL) were added to each tube in sequence; the contents of each tube were mixed evenly and placed in a 55°C oven for overnight. Next, 10M NH4OAC was added to the mixture in equal volume. The mixture was placed on ice for 5 minutes and centrifuged at 13,000 rpm for 10 minutes. The resulting supernatant was placed into a 1.5-mL centrifuge tube. Isopropanol was added to the resulting mixture in equal volume, and the mixture was stored at -20°C for overnight or -80°C for 1 hour. After centrifugation for 10 minutes at 13,000 rpm, the supernatants were removed from the precipitates, 75% alcohol (500µL) was added and left to stand for 5 minutes, and the mixture was centrifuged for 10 minutes at 13,000 rpm. The alcohol was then removed. Next, 100% alcohol (500µL) was added to the pellet. The mixture was left to stand for 5 minutes and subsequently centrifuged for 10 minutes at 13,000 rpm. Finally, the alcohol in the tube was poured out, and the centrifuge tube was placed upside down to allow any remaining alcohol to evaporate. Finally, the DNA precipitates were dissolved using an appropriate amount of sterilized water, placed into an oven at 55°C for 5 minutes, and stored at -20°C. Generally, the DNA specimens with an OD260/ OD280 ratio of 1.4 or higher. The concentration of recovered DNA was calculated on the basis of a concentration of 50 µg/mL at OD260 = 1.00, which was determined to be suitable for estimating the TOBC of each sample after the DNA quantification. Staphylococcus aureus (ATCC 29213) was used as the reference strain in bacterial growth curve estimation. After overnight culturing, the bacterial solution was serially diluted five times to generate specimens with different concentrations of S. aureus. A total of 10 µL of each of the specimens were taken and spread on the agar medium to attain concentrations of 2.5 × 103 to 3.9 × 107 CFU/mL. A volume of 1 mL of each different bacterial concentration was taken for bacterial DNA extraction. The extracted bacterial genomic DNA was stored frozen at -80°C until the RT-PCR test was conducted. Before the RT-PCR test, the bacterial genomic DNA concentration was measured. RT-PCR tests mainly detect 16S rRNA, and a StepOnePlus system (Applied Biosystems, Foster City, CA, USA) was used to establish a standard curve of S. aureus concentration. The sequence of the forward primer and reverse primer used were 5'-CCT ACG GGA GGC AGC AG-3' and 5'-CCG TCA ATT CMT TTR AGTT T-3', respectively.16 The coverage rates of selected forward and reverse primer pair for common bacterial species are 94.9% and 92.8%, respectively.16 The total PCR volume was 25 uL, comprising 5.5 µL of ddH2O, 1.0 µL of 5-µM preprimer, 1.0 µL of 5-µM reverse primer, 12.5 µL of SYBR solution, and 5.0 µL (0.25 µg) of DNA. The RT-PCR reaction conditions were as follows: 94°C for 10 minutes; followed by 35 cycles of 95°C for 45 seconds, 58°C for 40 seconds, and 72°C for 60 seconds; and followed by one cycle of 72°C for 7 minutes. A regression equation derived from the standard curve and the RT-PCR results were used to calculate the bacterial concentration in each saliva sample. The RT-PCR assay was conducted two duplicates for each sample, and the coefficient of variation of the threshold was varied between 2% and 12%. Human blood DNA was used as a negative control group.

Antibacterial activity of the mouthwash solution: The pure-cultured S. aureus used as the standard strain was plated on a culture plate (10 cm in diameter) containing 1.5% (g/L) luria broth agar and cultured overnight. A single colony was selected and placed in a conical flask containing LB nutrient liquid, shaken, and recultured overnight, and the resulting solution was serially diluted and coated on the plate to calculate the number of bacteria per unit volume. Finally, a Cell Counting Kit 8 (CCK-8, Engreen Biosystem) commercial reagent was used to evaluate the antibacterial effect of the mouthwash. Each experiment was performed in duplicate. Solutions containing different colony forming units (0, 10, 100, 1000, 10000, 100000, and 1000000) of S. aureus were centrifuged at 2000 rpm for 5 minutes to concentrate the bacteria; after the liquid was removed, 180 µL of fresh culture medium was added to suspend the bacteria in the culture medium. The bacteria solution was transferred to a 96-well plate. To evaluate the antibacterial effect of the mouthwash, 20 µL of the mouthwash was added to the mixture of the bacterial solution. The mixture was incubated at 37°C for 2 hours. Finally, 10 µL of CCK-8 reagent was added and mixed well. The resulting mixture was incubated at 37°C for 2 hours, and the absorbance at 450 nm was measured using an ELISA reader. The standard growth curve could be established for the estimation of the number of bacteria in the mixture and their survival rate of the bacteria, which were then compared with the standard curve.

Statistical analysis: After the data collection and checking were complete, the finalized debugged files were transferred to a computer with statistical software for statistical analysis. The descriptive statistics used included frequency distribution tables, percentages, means, and standard deviations. In the TOBC analysis, in addition to descriptive statistics, a t test, chi-square test, and linear regression analysis were conducted to assess and compare the changes in the bacterial counts of the participants' saliva after the intervention period. Considering the small sample size and the distribution of TOBC, nonparametric statistical methods were used for analysis. The Wilcoxon rank-sum test was used to identify differences in the numerical data of the intervention group and the control group, the Wilcoxon signed-rank test was used to identify changes in numerical data between the baseline and post-intervention, and the Kruskal-Wallis test and a post hoc Tukey test were used to identify differences in numerical data of three or more groups.

ELIGIBILITY:
Inclusion Criteria:

1. All the participants were between 35 and 70 years old.
2. Clinical diagnosis of periodontal disease
3. Must be able to rinse liquid (mouthwash or water) in mouth and split out saliva into a collection tube

Exclusion Criteria:

1. diagnosed mental illness
2. incapacitated patients
3. antibiotics or immunosuppressive drugs taken for the two consecutive weeks preceding study commencement
4. pregnant
5. smokers
6. cancers
7. Insulin dependent diabetes

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Total oral bacterial count before the intervention | Before the intervention starting
  Before the intervention, saliva samples were collected for oral bacterial DNA extraction.The saliva volume and weight of each sample was also recorded before the bacterial genomic DNA extraction process. A real-time polymerase chain reaction and S. aureus with serial dilutions were applied for the estimation of total oral bacterial count (TOBC) in saliva. The differences in TOBC among the mouthwash group (MW), mouthwash and periodontal flosser group (MWF), and control group were determined using statistical analysis.
Total oral bacterial count after the intervention | Immediately after the intervention
  After the intervention, saliva samples were collected for oral bacterial DNA extraction. The saliva volume and weight of each sample was also recorded before the bacterial genomic DNA extraction process. A real-time polymerase chain reaction and S. aureus with serial dilutions were applied for the estimation of total oral bacterial count (TOBC) in saliva. The difference in TOBC between before and after intervention was determined using statistical analysis
Survival rate of S. aureus after the incubation with 10% (v/v) mouthwash | One week after the intervention
  An in vitro assay and CCK-8 reagent were applied to determine the survival rates of 1000000 and 10000000 CFU/mL of S. aureus after being incubated with 10% (v/v) mouthwash. These results could indicate the anti-bacterial ability of mouthwash to S. aureus.

SECONDARY OUTCOMES:
The percentage change in the TOBC after the intervention | One month after the intervention
  The percentage change ((TOBC after intervention - TOBC before intervention)/ TOBC before intervention)*100%) in the TOBC of the MW, MWF, and control groups was determined after the intervention. Further to normalize the TOBC data by base-2 log-transformation, the change of TOBC were also determined after the intervention. Finally, the linear regression analysis was applied to determine the risk factors which could significantly affect the percentage change in TOBC after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hsian-Ling Huang, Ph.D., Principal Investigator — Kaohsiung Medical University; Ying-Chu Lin, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Private Wenhsin Dental Clinic, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin YC, Tsai CF, Huang HL. Effects of hypochlorous acid mouthwash on salivary bacteria including Staphylococcus aureus in patients with periodontal disease: a randomized controlled trial. BMC Oral Health. 2023 Sep 28;23(1):698. doi: 10.1186/s12903-023-03358-4. PMID 37770865